CLINICAL TRIAL: NCT07353905
Title: Intravascular Ultrasound Imaging Guidance for Optimal Revascularization of Limb Arteries
Acronym: INVIGOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 025-412
Record Dates: First submitted 2025-12-09; First posted 2026-01-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Arterial Disease; Femoropopliteal Disease
Keywords: Peripheral Artery Disease; Intravascular Ultrasound; Angioplasty; Endovascular Treatment
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Ultrasonography, Interventional

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled study.
Who Masked: Participant
Masking Description: Single-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intravascular Ultrasound (IVUS) (Active Comparator): Intravascular Ultrasound (IVUS) is used during the treatment of the target lesion.
  Interventions: Device: Intravascular Ultrasound (IVUS)
- Non-Intravascular Ultrasound (IVUS) (Active Comparator): Intravascular Ultrasound (IVUS) is not used in the treatment of the target lesion.
  Interventions: Device: Angiographic-guided Intervention

INTERVENTIONS:
Device: Intravascular Ultrasound (IVUS) — pre-and post-procedural IVUS to guide atherectomy, balloon angioplasty based treatments and/or stent placement
  Arms: Intravascular Ultrasound (IVUS)
Device: Angiographic-guided Intervention — Standard angiography-guided intervention without IVUS.
  Arms: Non-Intravascular Ultrasound (IVUS)

SUMMARY:
This study will test whether using ultrasound imaging within blood vessels during minimally invasive treatment of leg arteries in patients with peripheral artery disease leads to better clinical outcomes.

DETAILED DESCRIPTION:
This is a U.S. prospective multicenter randomized controlled trial to evaluate the clinical outcomes of Intravascular ultrasound (IVUS) guided Femoropopliteal (FP) endovascular intervention in patients with symptomatic peripheral artery disease (PAD) (Rutherford class 2-5).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years
* Symptomatic FP PAD with angiographic evidence of >50% stenosis
* Candidates for endovascular therapy

Exclusion Criteria:

* Prior intervention at the target lesion within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Primary Patency | From enrollment to 6 months
  Freedom from restenosis ≥50% or an increase in Duplex Ultrasound peak systolic velocity ≥2.5 times reference proximal segment or target lesion revascularization (TLR).

SECONDARY OUTCOMES:
Technical Success | Collected from index procedure
  Technical success is defined as less than 30% residual stenosis in the target lesion following the index procedure. Residual stenosis determined by operator visual estimation.
Procedural Success | Collected from Index procedure
  Procedural success is technical success (less than 30 % residual stenosis in the target lesion) without the occurrence of procedural complications during the index procedure. Residual stenosis determined by operator visual estimation.
Clinically driven-TLR (CD-TLR) | From enrollment to 12 months
  Clinically driven-target limb revascularization. Information collected from the medical record.
Amputation-free Survival | From enrollment to 12 months
  Defined as no evidence of amputation. Information is collected from the medical record
Functional Status Improvement (Vascular Quality of Life Questionnaire (VascuQoL-6)) | From enrollment to 12 months
  Vascular Quality of Life Questionnaire (VascuQoL-6) collected at index procedure and 12 months.
Functional Status Improvement (Rutherford Class Improvement) | From enrollment to 12 months
  Rutherford class determined by physician and collected from the medical record.
Cost Effectiveness | Evaluated at 12 months
  This analysis will calculate total cost-effectiveness by comparing costs between the two groups. Total cost will include the initial procedural cost, costs related to complications, and costs of any repeat reinterventions during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Subhash Banerjee, MD, Principal Investigator — Baylor Scott & White Research Institute
Locations (6):
- United States (6):
  - Baylor Scott & White The Heart Hospital - Dallas, Dallas, Texas
  - Baylor Scott & White The Heart Hospital - Fort Worth, Fort Worth, Texas
  - Baylor Scott & White The Heart Hospital - Mckinney, McKinney, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Baylor Scott & White Medical Center - Temple, Temple, Texas
  - Baylor Scott & White The Heart Hospital - Waxahachie, Waxahachie, Texas

IPD SHARING:
Plan to Share IPD: No
We will need to get Information Security and sponsor approval before sharing our data. Any data shared would be aggregate, de-identified data shared in accordance with Baylor Scott & White Research Institute's policies and procedures.

REFERENCES:
- [Result] Jang JS, Jin HY, Park YA, Yang TH, Seo JS, Kim DK, Wi JH. Meta-Analysis of Intravascular Ultrasound-Guided Versus Angiography-Guided Endovascular Treatment in Lower Extremity Artery Disease. Am J Cardiol. 2025 Mar 15;239:8-17. doi: 10.1016/j.amjcard.2024.12.012. Epub 2024 Dec 12. PMID 39674438
- [Result] Secemsky EA, Aronow HD, Kwolek CJ, Meissner M, Muck PE, Parikh SA, Winokur RS, George JC, Salazar G, Murphy EH, Costantino MM, Zhou W, Li J, Lookstein R, Desai KR. Intravascular Ultrasound Use in Peripheral Arterial and Deep Venous Interventions: Multidisciplinary Expert Opinion From SCAI/AVF/AVLS/SIR/SVM/SVS. J Vasc Interv Radiol. 2024 Mar;35(3):335-348. doi: 10.1016/j.jvir.2023.11.006. Epub 2024 Jan 9. PMID 38206255
- [Result] Korosoglou G, Schmidt A, Lichtenberg M, Malyar N, Stavroulakis K, Reinecke H, Grozinger G, Patrone L, Varcoe RL, Soukas PA, Bockler D, Behrendt CA, Secemsky EA, Zeller T, Blessing E, Langhoff R, Rammos C. Global Algorithm for the Endovascular Treatment of Chronic Femoropopliteal Lesions: An Interdisciplinary Expert Opinion Statement. JACC Cardiovasc Interv. 2025 Mar 10;18(5):545-557. doi: 10.1016/j.jcin.2024.11.038. PMID 40074516
- [Result] Halabi S, Al Hennawi H, Secemsky EA, Palena M, Manzi M. Intravascular Ultrasound Guided Puncture of Stumpless Tibial Occlusions. Am J Cardiol. 2025 Nov 1;254:108-112. doi: 10.1016/j.amjcard.2025.08.002. Epub 2025 Aug 9. PMID 40789536
- [Result] Lee SJ, Kim TH, Lee JH, Ahn CM, Lee SH, Lee YJ, Kim BK, Hong MK, Jang Y, Park HW, Jang JY, Park JH, Kim SH, Im E, Park SH, Choi D, Ko YG; IVUS-DCB Investigators. Intravascular Ultrasound-Guided vs Angiography-Guided Drug-Coated Balloon Angioplasty in Patients With Complex Femoropopliteal Artery Disease. JACC Cardiovasc Interv. 2025 Mar 10;18(5):558-569. doi: 10.1016/j.jcin.2024.10.052. Epub 2025 Jan 22. PMID 39846915
- [Result] Soney H, Kakkilaya A, Vazquez DF, Banerjee R, Rosol Z, Tsai S, Banerjee S. Reproducibility of Femoropopliteal Artery Intravascular Ultrasound Imaging in Patients With Peripheral Artery Disease. Am J Cardiol. 2023 Jul 15;199:1-6. doi: 10.1016/j.amjcard.2023.04.026. Epub 2023 May 19. PMID 37210800

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-02-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT07353905/Prot_SAP_001.pdf